CLINICAL TRIAL: NCT06253598
Title: Efficacy and Safety of Intratumoral Injection of Recombinant Human Adenovirus Type 5 Combined With Tislelizumab and Lenvatinib in the Treatment of Advanced Hepatocellular Carcinoma: a Single-center, Prospective, Single-arm Study
Brief Title: Efficacy and Safety of Intratumoral Injection of Recombinant Human Adenovirus Type 5 Combined With Tislelizumab and Lenvatinib in the Treatment of Advanced Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital of Bengbu Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCC-01
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-02

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — lenvatinib; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- intervention arm (Experimental)
  Interventions: Drug: Recombinant Human Adenovirus Type 5; Drug: Lenvatinib; Drug: Tislelizumab

INTERVENTIONS:
Drug: Recombinant Human Adenovirus Type 5 — Recombinant Human Adenovirus Type 5( H101 )was administered intratumorally on day 1 and 5 of cycle 1 and cycle 2. If the sum of the maximum diameters of the lesions was less than or equal to 10 cm, the total dose was 1.0×10^12 vp . If the sum of the maximum diameters of the lesions was more than 10 cm, the total dose was 1.5×10^12 vp. Recombinant Human Adenovirus Type 5 was diluted to 30% of the total tumor volume with normal saline before administration. Under the guidance of ultrasound, percutaneous puncture was performed to the center of the tumor, and the solution was uniformly injected into the tumor. If there are multiple lesions, the distribution of each lesion should be proportional to the size of the tumor. No more than 5 lesions.
  Other Names: H101
Drug: Lenvatinib — Lenvatinib was administered orally once daily started on day 1 of cycle 1 of the study until disease progression or unacceptable toxicity occurred or meet the end point of the study. For patients weighing less than 60 kg, the recommended daily dose was 8 mg once daily. For patients weighing ≥60 kg, the recommended daily dose was 12 mg once daily
Drug: Tislelizumab — Tislelizumab 200mg was administered intravenously every 3 week started on day 1 of cycle 3 until disease progression or unacceptable toxicity occurred or meet the end point of the study.

SUMMARY:
This prospective, single-arm study was aimed to evaluate the efficacy of recombinant human adenovirus type 5 injection combined with tislelizumab and lenvatinib in the treatment of advanced hepatocellular carcinoma. The recombinant human adenovirus type 5 was administered intratumorally on day 1 and 5 in cycle 1 and cycle 2. Lenvatinib was administered orally once daily started on day 1 of cycle 1 .Tislelizumab was administered intravenously every 3 week started on day 1 of cycle 3. The patient accepted the therapy until disease progression or unacceptable toxicity occurred or meet the end point of the study. The primary end point was ORR assessed by investigator using RECIST v1.1 .

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years old, and ≤75 years old, regardless of gender;
2. Primary hepatocellular carcinoma confirmed by histology or imaging;
3. Patients with advanced hepatocellular carcinoma who have not received oncolytic viruses, immutherapy drugs (including anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs), and systemic therapy (such as anti-VEGF /VEGFR monoclonal antibodies, anti- VEGFR-TKI drugs, chemotherapy);
4. ECOG performance status 0-1;
5. Child-Pugh score ≤7;
6. There was at least one measurable target lesion according to RECIST 1.1 criteria, and at least one lesion was ≥ 10 mm;
7. The expected survival time was ≥3 months;
8. Laboratory tests during the screening period met the following criteria:

   i. White blood cell count ≥ 3.0×10^9 /L, absolute neutrophil count ≥1.5×10^9/L, platelet count ≥ 75×10^9/L, hemoglobin > 90g/L

   ii. INR≤1.5 and APTT≤1.5 times upper limit of normal or partial prothrombin time (PTT) ≤1.5 times upper limit of normal;

   iii. Total bilirubin ≤2.5 times upper limit of normal; ALT and AST≤5 times upper limit of normal (ULN); Serum creatinine ≤1.5 times the upper limit of normal.
9. They volunteered to participate in this study and signed informed consent.

Exclusion Criteria:

1. Pregnant or lactating women, men or women unwilling to use effective contraception;
2. Diffuse liver cancer or tumor is not suitable for RECIST 1.1 criteria;
3. Patients who have previously received an oncolytic viral agent such as T-VEC;
4. Known allergy to the study drug or its active ingredient, history of allergy to the same biological agent;
5. HBV DNA quantitation ≥1000 copies.
6. Imaging showed portal vein tumor thrombus more than half of the lumen, inferior vena cava tumor thrombus or heart involvement.
7. The patient has had grade ≥2 hepatic encephalopathy within 12 months or currently requires medication to prevent or control hepatic encephalopathy.
8. Confirmed active tuberculosis (TB), known human immunodeficiency virus (HIV) positive patients, and other serious infections requiring treatment;
9. A history of immunodeficiency or autoimmune disease, or long-term systemic steroid therapy or any form of immunosuppressive therapy within 7 days before enrollment;
10. A history of other (including unknown primary) malignancies, except for Cured non- melanoma skin malignancies, carcinoma in situ of the cervix, radical stage I uterine cancer, radical ductal carcinoma in situ or lobular carcinoma in situ of the breast (without any systemic treatment), localized prostate cancer that is currently considered cured after radical surgery, and other solid tumors that have been treated with radical surgery for more than 5 years without evidence of recurrence;
11. Known tumors of the central nervous system, including metastatic brain tumors;
12. Accompanied by any unstable systemic disease, including but not limited to: Severe infections, patients with hypertension whose blood pressure cannot be lowered to normal after antihypertensive treatment, uncontrolled diabetes mellitus, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, myocardial infarction (a history of myocardial infarction of 6 months or more is allowed), congestive heart failure, serious arrhythmias requiring medical treatment, renal or metabolic diseases;
13. With medical contraindications to any contrast-enhanced imaging (CT or MRI);
14. Participants who had participated in an interventional clinical trial within 30 days before screening (Note: Participants who were already in the follow-up phase of the clinical trial could participate in this trial if it was 4 weeks after the last dose of the previous investigational drug).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-03-30 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Objective response rate using RECIST v1.1 | 3 years
  ORR is defined as the proportion of patients who have a partial or complete response to therapy

SECONDARY OUTCOMES:
DOT | 3 years
  Duration of treatment
DOR | 3 years
  Duration of response
DCR | 3 years
  Disease control rate
PFS | 3 years
  progression-free survival
1-year overall survival rate | 1years
  the overall survival rate at 1 year
AE | 3 years
  adverse events base on CTCAE v5.0

IPD SHARING:
Plan to Share IPD: No